CLINICAL TRIAL: NCT02917889
Title: Acute Caffeine Effects on Cardiac Autonomic and Cardiorespiratory Parameters Responses After Aerobic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luana Almeida Gonzaga, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 44888015.8.0000.5406
Record Dates: First submitted 2016-09-19; First posted 2016-09-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Autonomic Nervous System; Cardiorespiratory Parameters
Keywords: Caffeine; Autonomic Nervous System; Recovery; Aerobic exercise
MeSH Terms: interventions — Caffeine; Exercise Test

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Caffeine protocol (Experimental): 300 mg in pills
  Interventions: Drug: Caffeine; Other: Cardiopulmonary test; Other: Treadmill aerobic exercise
- Placebo protocol (Experimental): 300 mg in pills
  Interventions: Drug: Placebo; Other: Cardiopulmonary test; Other: Treadmill aerobic exercise

INTERVENTIONS:
Drug: Caffeine — Volunteers will consume 300 mg of caffeine in pills fifteen minutes before treadmill aerobic exercise.
  Arms: Caffeine protocol
Drug: Placebo — Volunteers will consume 300 mg of placebo in pills fifteen minutes before treadmill aerobic exercise.
  Arms: Placebo protocol
Other: Cardiopulmonary test — assessment of the maximum oxygen consumption (VO2max) on a treadmill (Inbrasport / Millennium), using Buce protocol.
  .
Other: Treadmill aerobic exercise — 30 mim of aerobic exercise (5 minutes at speed of 5.0 km/h for warming-up followed by 25 minutes at 60% of VO2max ).

SUMMARY:
Check the acute influence of caffeine on the autonomic modulation and cardiorespiratory parameters after aerobic exercise. Hypothesized that caffeine can promote a slower recovery of the cardiorespiratory parameters and the SNA recovery after aerobic exercise.

DETAILED DESCRIPTION:
The experimental procedure is divided into three phases, all performed on a treadmill, with a minimum interval of 48 hours between them, in order to allow adequate recovery of the participants. Before the start of the first stage of the experimental protocol or control anthropometric measurements will be carried out, body weight by a digital scale (Plenna, TIN 00139 MAXIMA, Brazil)) and then, using a stadiometer (Plenna, TIN 00139 MAXIMA, Brazil)). The protocols are:

I) Maximum stress test protocol: assessment of the maximum oxygen consumption (VO2max) on a treadmill (Inbrasport / Millennium), using the Bruce protocol.

II) Control Protocol (PC): at this stage the volunteer will ingest compressed form of placebo similar to Protocol III and remained at rest after 15 minutes in the supine position, followed by 30 minutes of aerobic exercise on a treadmill, 5 minutes with speed 6.0 km / h followed by 25 minutes with 60% of VO2max and the final 60 minutes lying recovery.

III) Experimental protocol (PE): In this stage, the volunteer had performed activities similar to the PC, but will make the tablet intake consists of 300mg of caffeine, a value that is within the maximum daily amount allowed under the FDA.

ELIGIBILITY:
Inclusion Criteria:

* healthy men.

Exclusion Criteria:

* cardiovascular, orthopedic, respiratory and neurological disorders reported or other pathological conditions that prevent the subject to perform the protocols;
* smokers, alcoholics, or who use drugs that influence the activity of the heart.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Caffeine effects on heart rate variability (based on frequency, time domain and Chaos) | up to 1 year
Blood pressure (mmHg) | up to 1 year
  Caffeine effects blood pressure recovery following aerobic exercise
Heart rate (beats per minute) | up to 1 year
  Caffeine effects heart rate recovery following aerobic exercise
Respiratory rate (per minute) | up to 1 year
  Caffeine effects arespiratory rate recovery following aerobic exercise
Oxygen saturation pulse (oximeter-SpO2) | up to 1 year
  Caffeine effects SpO2 recovery following aerobic exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual Paulista, Presidente Prudente, São Paulo, Brazil